CLINICAL TRIAL: NCT05783856
Title: Application of Vaginal-spraying LiveSpo X-secret in Supporting Treatment of Sexually Transmitted Diseases in Vietnamese Women
Brief Title: Effects of LiveSpo X-secret in Supporting Treatment of Sexually Transmitted Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Hanoi University of Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-1906
Record Dates: First submitted 2023-03-11; First posted 2023-03-24 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Sexually Transmitted Diseases
Keywords: Sexually Transmitted Diseases (STDs); Sexually Transmitted Infections (STIs); Bacterial vaginosis (BV); Vaginal-spraying probiotics; Bacillus spores; Pathogen load; Fungi; Virus; Vietnamese women
MeSH Terms: conditions — Sexually Transmitted Diseases; Vaginosis, Bacterial; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo X-secret and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo X-secret suspension is unrecognizable to investigators except the PI and analyzer due to opaque plastic container
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control group receives the routine treatment and uses 0.9% NaCl physiological saline.
  The routine treatment regimen at the Bac Ninh Center for Disease Control depends on the type of pathogen tested using multiplex real time PCR assay on day 0, as follows:
  Oral administrative medication based on the results of STIs pathogen detection test, antibiotic Clinidamycin (Withus Clinidamycin®) or/and the antifungal drug Itraconazole (Miduc®) are prescribed for 7 days to treat pathogenic bacteria or/and fungi infections, respectively.
  Vaginal suppository medication: Canvey®, which contains Metronidazole and Chloramphenicol, is only prescribed for further 7 days in the event that oral treatments of Clindamycin and Itraconazole have been unsuccessful.
  Interventions: Drug: 0.9% NaCl physiological saline
- X-secret (Experimental): X-secret group receives the routine treatment and uses NaCl 0.9% plus B. subtilis, B. clausii, and B. coagulans at 5 billion CFU/5 mL (LiveSpo®️ X-secret).
  The routine treatment regimen at the Bac Ninh Center for Disease Control depends on the type of pathogen tested using multiplex real time PCR assay on day 0, as follows:
  Oral administrative medication based on the results of STIs pathogen detection test, antibiotic Clinidamycin (Withus Clinidamycin®) or/and the antifungal drug Itraconazole (Miduc®) are prescribed for 7 days to treat pathogenic bacteria or/and fungi infections, respectively.
  Vaginal suppository medication: Canvey®, which contains Metronidazole and Chloramphenicol, is only prescribed for further 7 days in the event that oral treatments of Clindamycin and Itraconazole have been unsuccessful.
  Interventions: Combination Product: LiveSpo X-secret

INTERVENTIONS:
Combination Product: LiveSpo X-secret — In Vietnam, LiveSpo X-secret is manufactured as a Class-A medical device product (Product declaration No.220003286/PCBA-HN) under manufacturing standards approved by Hanoi Health Department, Ministry of Health, Vietnam (Certificate No YT117-19) and ISO 13485:2016.
  Other Names: Registration number: No.220003286/PCBA-HN
  Arms: X-secret
Drug: 0.9% NaCl physiological saline — Vaginal-spraying 0.9% NaCl physiological saline is prepared by extracting 10 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque metallic spraying 15 mL-bottle that is used for LiveSpo X-secret.
  Other Names: Registration number: VD-32723-19
  Arms: Control

SUMMARY:
Sexually Transmitted Infections (STIs) are common gynecological infections worldwide, especially in tropical and underdeveloped countries, primarily affecting the reproductive age group. Microbial pathogens causing STIs include bacteria, viruses, fungi, and protozoa. In Vietnam, STIs are a significant public health concern due to their high incidence and tendency to have mild or no symptoms, making them easy to overlook. While antibiotics or antifungal drugs are typically used to treat STIs caused by bacterial or fungal agents such as Chlamydia, Gonorrhea, and Candida, no specific treatment exists for most viral STIs. Thus, vaccination and symptomatic treatment are the primary methods of prevention. The use of broad-spectrum antibiotics can result in side effects such as loss of appetite, fatigue, and sexual problems, while repeated treatments can lead to the emergence of antibiotic resistance, posing a significant challenge for STI treatment worldwide. However, the efficacy of oral or suppository-based probiotics is limited by their slow onset and sensitivity to acidic and temperature conditions. Fortunately, Bacillus strains of probiotics have demonstrated exceptional stability in both acidic and temperature environments, making them particularly well-suited for use as vaginal spray probiotics against STIs. Here, investigators propose that vaginal-spraying probiotics containing Bacillus strains could be a safe and effective symptomatic treatment for STIs caused by viral, fungi, or bacterial pathogens, providing a promising alternative to traditional antibiotic therapy.

The aim of the study about to evaluate the effectiveness of vaginal-spraying probiotics containing spores of three strains of Bacillus subtilis, Bacillus clausii, and Bacillus coagulans in preventing and supporting the treatment of vaginal infections.

Study Population: sample size is 100. The study is being carried out at Bac Ninh Center for Disease Control.

Description of Study Intervention: total of 100 eligible patients are divided randomly into 2 groups (n = 50/group): Patients in the Control group received routine treatment and 3 times/day 0.9% NaCl physiological saline while the patients in the experimental group were treated with LiveSpo X-secret 3 times/day in addition to the same standard of care treatment. The standard treatment regimen is 7 days and is maintained for 28 days.

Study duration: 36 months

DETAILED DESCRIPTION:
Sexually Transmitted Infections (STIs) are common gynecological infections worldwide, especially in tropical and underdeveloped countries where up to three-quarters of the population has STIs, mainly in the reproductive age. The infection rate in regions and countries is different, the infection rate in developing countries is 20-fold higher than in developed countries. Southeast Asia alone has about 150.5 million people with these diseases. Vietnam is located in the tropics, and hot and humid climates are favorable factors for microbial pathogens to develop. According to reports from the dermatology units of the provinces, every year about 300,000 people are infected with sexually transmitted diseases...There are many microbial pathogens causing infections including bacteria, viruses, fungi, and protozoa...The patient can be infected with multiple pathogens at the same time. This is a matter of great concern in public health care because STIs often have mild or no symptoms, so they are easily overlooked. While antibiotics or antifungal drugs are typically used to treat STIs caused by bacterial or fungal agents like Chlamydia, Gonorrhea, and Candida, no specific treatment exists for most viral STIs. However, the use of broad-spectrum antibiotics can result in side effects like loss of appetite, fatigue, and sexual problems, while repeated treatments can lead to the emergence of antibiotic resistance, posing a significant challenge for STI treatment worldwide. Probiotics are microorganisms that are beneficial to our health when consumed in adequate amounts, playing a vital role in maintaining a healthy balance of bacteria in our body, especially in the gut and vaginal areas. Studies have found that probiotics can help reduce the incidence and severity of vaginal infections, including bacterial vaginosis and yeast infections. Currently, oral or vaginal suppository probiotics containing strains of Bifidobacterium or Lactobacillus are being studied as a potential complementary therapy for treating vaginal infections. However, these strains have low survivability and are sensitive to light, moisture, and pH levels, making preservation challenging. Thus, their effectiveness depends on the specific strains used and the dose required to achieve colonization in the vaginal tract. Bacillus is a well-studied probiotic strain with over 350,000 research publications worldwide, and its safety has been extensively investigated. Bacillus subtilis, B. clausii, and B. coagulans are all aerobic or facultative anaerobic bacteria capable of spore formation and can tolerate harsh conditions such as nutrient deprivation, anoxia, drought, and even antibiotics. Here, investigators propose that vaginal-spraying probiotics containing Bacillus strains could be a safe and effective symptomatic treatment for STIs caused by viral, fungi, or bacterial pathogens, providing a promising alternative to traditional antibiotic therapy.

The objective was to investigate the symptomatic treatment effects of the probiotic product LiveSpo X-secret as a liquid-suspension form containing Bacillus spores of safe B. subtilis ANA4, B. clausii ANA39, B. coagulans ANA 40 strains, in women having sexually transmitted infection and investigators evaluation of improved efficacy and reduced clinical symptoms treatment time and measurement of changes in pathogen load in the vaginal samples before treatment (day 0) and after 3, 7, 14 and 28 days using LiveSpo X-secret.

Methods: A randomized, blind, and controlled clinical trial is conducted. After informed consent, patients will be screened for common nine STI pathogens in Vietnam including Gardnerella vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Mycoplasma hominis, Mycoplasma genitalium, Human alphaherpesvirus type 1 and 2, Candida albicans, Trichomonas vaginalis. Totally 100 patients positive with at least one of nine STIs will be randomized into 2 groups (n = 50/group): the control group (named "Control" group) uses 0.9% NaCl physiological saline and an experimental group (named the "X-secret" group) use the probiotics LiveSpo X-secret. The patient is given a coded spray in the form of a blind sample to ensure the objectivity of the study. The clinical follow-up will be at the time point of 0, 3, 7, 14, and 28 days, vaginal samples will be collected at days 0, 3, 7, 14, and day 28 to evaluate potential reductions in pathogens load and change the microbiome in vaginal flora.

Real-time PCR for detection of microorganism in vaginal samples: semi-quantitative assays for measuring changes in pathogens load is conducted by the real-time PCR assay which has been optimized and developed by the research team (Bui et al., 2023). Detection of useful Bacillus strains belonging to B. subtilis, B. clausii, and B. coagulans is conducted by real-time PCR SYBR Green assay that is routinely runs also conducted at Spobiotic Research Center, Hanoi, Vietnam

Analysis of vaginal microbiome 16S rRNA using next-generation sequencing (NGS) at Macrogene (Seoul, Korea) on the Illumina MiSeq (Illumina, San Diego, CA, USA) using a 2 × 250 bp run configuration.

During treatment, patients are monitored for typical clinical symptoms of gynecological infections, including itching, odor, vaginal color, and pH from vaginal samples of Control and X-secret groups at the time points of day 3, 7, 14, and day 28. The patients' health conditions are observed by doctors and nurses, and their pieces of information are filled into medical records at the patient's follow-up visits or phone interviews.

Data collection and statistical analysis: individual medical records are collected, and the patient's information is then gathered and systematized in a data set. The safety and efficacy of LiveSpo X-secret are evaluated and compared to 0.9% NaCl physiological saline based on the following clinical and sub-clinical criteria obtained in X-secret and Control groups: (i) the symptomatic-relieving day and level of symptom relief; (ii) the reduction levels (2^△Ct) of pathogens load △Ct for target genes is calculated as Ct (threshold cycle) at day 3/7/14/28 - Ct at day 0 while Ct of internal control is adjusted to be equal among all samples; (iii) change the microbiome in vaginal flora.

The tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using either the Wilcoxon test, t-test, or the Mann-Whitney test when data are not normally distributed. Statistical and graphical analyses are performed on GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level of all analyses is set at p < 0.05. P-values.

Expected outcomes: (i) LiveSpo X-secret alleviates influenza-infection symptoms about 30% more effectively, as indicated by 90% of patients using LiveSpo X-secret (X-secret group) are symptom-free at day 3-28 of intervention depending on symptoms, compared to 60% of patients in Control group; (ii) Patients in X-secret group has more significant reductions in pathogens load (>10 fold) than patients in Control group at the time point of day 3, 7, 14, 28 of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18 to 60 years
* Amsel criteria for the diagnosis of vaginitis (presence of 3 of the following four criteria)

  * Increased uniform thin vaginal discharge;
  * pH of vaginal discharge greater than 4.5;
  * Vaginal odor;
* STI positive detected by multiplex real-time PCR TaqMan probe for nine major vaginal pathogens circulating in Vietnam. These include Gardnerella vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Mycoplasma hominis, Mycoplasma genitalium, Human alphaherpesvirus type 1 and 2, Candida albicans, Trichomonas vaginalis;
* Patients agree to participate in the study after a thorough explanation of the research is provided to them, and they sign the research consent form.

Exclusion Criteria:

* Pregnant or nursing women, diabetics, taking antibiotics or antibiotics against vaginal infections in the previous 14 days.
* Unexplained vaginal bleeding or cancer.
* Having a history of drug allergies and hypersensitivity to any ingredient in probiotics or placebo.
* Discharged before day 7
* Meeting the criteria for psychiatric disorders other than depression and/or anxiety.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gynecological infections are related to the vaginal tract of women. We are currently testing on women.
Enrollment: 100 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with free and/or reduced gynecological infection symptoms | Day 0 to day 28
  Percentage of patients with free gynecological infection including itching, odor, vaginal color, painful urination/ burning urine and lower abdominal pain
  * Vaginal itching/ odor level (rating from 0 to 3 on a scale of: None-0, Mild-1, Severe-2, Very severe-3)
  * Colored vaginal discharge (Clear white-0, Opaque-1,Yellow/green-2, Gray white-3)
  * Painful urination/ burning urine (Yes/No)
  * Lower abdominal pain (Yes/No)

SECONDARY OUTCOMES:
Change the vaginal pathogens load | Day 0, 3, 7, 14, and day 28
  Change the concentration of pathogens in vaginal samples, as indicated by real-time PCR threshold cycle (Ct) value at day 3, day 7, day 14 and day 28 (after treatment) compared with day 0 (before treatment)
Change the vaginal pH values | Day 0, 3, 7, 14, and day 28
  Change the pH values of vaginal samples at day 3, day 7, day 14 and day 28 (after treatment) compared with day 0 (before treatment)
Change the vaginal flora | Day 0, 7, and day 28
  Change the microbiome in vaginal flora, as indicated by the diversity of vaginal microbial species based on the data analysis of next-generation sequencing (NGS) at day 7 and day 28 (after treatment) compared with day 0 (before treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Ha TV Bui, PhD., Principal Investigator — VNU University of Sciences, Viet Nam National University; Anh TV Nguyen, PhD., Principal Investigator — Spobio Research Center, ANABIO R&D Ltd., Hanoi, Vietnam
Locations (1):
- Bac Ninh Center of Disease Control, Bắc Ninh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study peport (CSR). For more information or to submit a request, please contact clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Background] Izetbegovic S, Alajbegovic J, Mutevelic A, Pasagic A, Masic I. Prevention of diseases in gynecology. Int J Prev Med. 2013 Dec;4(12):1347-58. PMID 24498489
- [Background] Garrett N, Mitchev N, Osman F, Naidoo J, Dorward J, Singh R, Ngobese H, Rompalo A, Mlisana K, Mindel A. Diagnostic accuracy of the Xpert CT/NG and OSOM Trichomonas Rapid assays for point-of-care STI testing among young women in South Africa: a cross-sectional study. BMJ Open. 2019 Feb 19;9(2):e026888. doi: 10.1136/bmjopen-2018-026888. PMID 30782948
- [Background] Van der Pol B. Trichomonas vaginalis infection: the most prevalent nonviral sexually transmitted infection receives the least public health attention. Clin Infect Dis. 2007 Jan 1;44(1):23-5. doi: 10.1086/509934. Epub 2006 Nov 27. No abstract available. PMID 17143810
- [Background] Bebear C, de Barbeyrac B. Genital Chlamydia trachomatis infections. Clin Microbiol Infect. 2009 Jan;15(1):4-10. doi: 10.1111/j.1469-0691.2008.02647.x. PMID 19220334
- [Background] Gavin L, MacKay AP, Brown K, Harrier S, Ventura SJ, Kann L, Rangel M, Berman S, Dittus P, Liddon N, Markowitz L, Sternberg M, Weinstock H, David-Ferdon C, Ryan G; Centers for Disease Control and Prevention (CDC). Sexual and reproductive health of persons aged 10-24 years - United States, 2002-2007. MMWR Surveill Summ. 2009 Jul 17;58(6):1-58. PMID 19609250
- [Background] Campos GB, Lobao TN, Selis NN, Amorim AT, Martins HB, Barbosa MS, Oliveira TH, dos Santos DB, Figueiredo TB, Miranda Marques L, Timenetsky J. Prevalence of Mycoplasma genitalium and Mycoplasma hominis in urogenital tract of Brazilian women. BMC Infect Dis. 2015 Feb 14;15:60. doi: 10.1186/s12879-015-0792-4. PMID 25886914
- [Background] Chesson HW, Mayaud P, Aral SO. Sexually Transmitted Infections: Impact and Cost-Effectiveness of Prevention. In: Holmes KK, Bertozzi S, Bloom BR, Jha P, editors. Major Infectious Diseases. 3rd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2017 Nov 3. Chapter 10. Available from http://www.ncbi.nlm.nih.gov/books/NBK525195/ PMID 30212101
- [Background] Denning DW, Kneale M, Sobel JD, Rautemaa-Richardson R. Global burden of recurrent vulvovaginal candidiasis: a systematic review. Lancet Infect Dis. 2018 Nov;18(11):e339-e347. doi: 10.1016/S1473-3099(18)30103-8. Epub 2018 Aug 2. PMID 30078662
- [Background] Paladine HL, Desai UA. Vaginitis: Diagnosis and Treatment. Am Fam Physician. 2018 Mar 1;97(5):321-329. PMID 29671516
- [Background] Bui HTV, Bui HT, Chu SV, Nguyen HT, Nguyen ATV, Truong PT, Dang TTH, Nguyen ATV. Simultaneous real-time PCR detection of nine prevalent sexually transmitted infections using a predesigned double-quenched TaqMan probe panel. PLoS One. 2023 Mar 6;18(3):e0282439. doi: 10.1371/journal.pone.0282439. eCollection 2023. PMID 36877694
- [Background] Pham QD, Nguyen TV, Hoang CQ, Cao V, Khuu NV, Phan HT, Mai AH, Tran HN, Wilson DP, Zhang L. Prevalence of HIV/STIs and associated factors among men who have sex with men in An Giang, Vietnam. Sex Transm Dis. 2012 Oct;39(10):799-806. doi: 10.1097/OLQ.0b013e318265b180. PMID 23001268
- [Background] Nguyen BH, Pham QM, Hoang L, Sansone A, Jannini EA, Tran CM. Investigating the microbial pathogens of sexually transmitted infections among heterosexual Vietnamese men with symptomatic urethritis. Aging Male. 2022 Dec;25(1):125-133. doi: 10.1080/13685538.2022.2063272. PMID 35416126
- [Background] Rowley J, Vander Hoorn S, Korenromp E, Low N, Unemo M, Abu-Raddad LJ, Chico RM, Smolak A, Newman L, Gottlieb S, Thwin SS, Broutet N, Taylor MM. Chlamydia, gonorrhoea, trichomoniasis and syphilis: global prevalence and incidence estimates, 2016. Bull World Health Organ. 2019 Aug 1;97(8):548-562P. doi: 10.2471/BLT.18.228486. Epub 2019 Jun 6. PMID 31384073
- [Background] Garcia MR, Leslie SW, Wray AA. Sexually Transmitted Infections. 2024 Apr 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560808/ PMID 32809643
- [Background] Kaur IP, Chopra K, Saini A. Probiotics: potential pharmaceutical applications. Eur J Pharm Sci. 2002 Feb;15(1):1-9. doi: 10.1016/s0928-0987(01)00209-3. PMID 11803126
- [Background] Mastromarino P, Vitali B, Mosca L. Bacterial vaginosis: a review on clinical trials with probiotics. New Microbiol. 2013 Jul;36(3):229-38. Epub 2013 Jun 30. PMID 23912864
- [Background] Falconi-McCahill A. Bacterial Vaginosis: A Clinical Update with a Focus on Complementary and Alternative Therapies. J Midwifery Womens Health. 2019 Sep;64(5):578-591. doi: 10.1111/jmwh.13013. Epub 2019 Aug 1. PMID 31368667
- [Background] Lee NK, Kim WS, Paik HD. Bacillus strains as human probiotics: characterization, safety, microbiome, and probiotic carrier. Food Sci Biotechnol. 2019 Oct 8;28(5):1297-1305. doi: 10.1007/s10068-019-00691-9. eCollection 2019 Oct. PMID 31695928
- [Background] Torres-Sanchez A, Pardo-Cacho J, Lopez-Moreno A, Ruiz-Moreno A, Cerk K, Aguilera M. Antimicrobial Effects of Potential Probiotics of Bacillus spp. Isolated from Human Microbiota: In Vitro and In Silico Methods. Microorganisms. 2021 Jul 29;9(8):1615. doi: 10.3390/microorganisms9081615. PMID 34442694
- [Background] Ma L, Su J, Su Y, Sun W, Zeng Z. Probiotics administered intravaginally as a complementary therapy combined with antibiotics for the treatment of bacterial vaginosis: a systematic review protocol. BMJ Open. 2017 Oct 15;7(10):e019301. doi: 10.1136/bmjopen-2017-019301. PMID 29038188
- [Background] Falagas ME, Betsi GI, Athanasiou S. Probiotics for prevention of recurrent vulvovaginal candidiasis: a review. J Antimicrob Chemother. 2006 Aug;58(2):266-72. doi: 10.1093/jac/dkl246. Epub 2006 Jun 21. PMID 16790461
- [Background] Petrova MI, Lievens E, Malik S, Imholz N, Lebeer S. Lactobacillus species as biomarkers and agents that can promote various aspects of vaginal health. Front Physiol. 2015 Mar 25;6:81. doi: 10.3389/fphys.2015.00081. eCollection 2015. PMID 25859220
- [Background] Parma M, Dindelli M, Caputo L, Redaelli A, Quaranta L, Candiani M. The role of vaginal Lactobacillus Rhamnosus (Normogin(R)) in preventing Bacterial Vaginosis in women with history of recurrences, undergoing surgical menopause: a prospective pilot study. Eur Rev Med Pharmacol Sci. 2013 May;17(10):1399-403. PMID 23740456
- [Background] Mastromarino P, Macchia S, Meggiorini L, Trinchieri V, Mosca L, Perluigi M, Midulla C. Effectiveness of Lactobacillus-containing vaginal tablets in the treatment of symptomatic bacterial vaginosis. Clin Microbiol Infect. 2009 Jan;15(1):67-74. doi: 10.1111/j.1469-0691.2008.02112.x. Epub 2008 Nov 22. PMID 19046169
- [Background] Reid G, Charbonneau D, Erb J, Kochanowski B, Beuerman D, Poehner R, Bruce AW. Oral use of Lactobacillus rhamnosus GR-1 and L. fermentum RC-14 significantly alters vaginal flora: randomized, placebo-controlled trial in 64 healthy women. FEMS Immunol Med Microbiol. 2003 Mar 20;35(2):131-4. doi: 10.1016/S0928-8244(02)00465-0. PMID 12628548
- [Background] Hemalatha R, Mastromarino P, Ramalaxmi BA, Balakrishna NV, Sesikeran B. Effectiveness of vaginal tablets containing lactobacilli versus pH tablets on vaginal health and inflammatory cytokines: a randomized, double-blind study. Eur J Clin Microbiol Infect Dis. 2012 Nov;31(11):3097-105. doi: 10.1007/s10096-012-1671-1. Epub 2012 Jul 10. PMID 22777592
- See also: Sexually transmitted infections (STIs) — https://www.who.int/news-room/fact-sheets/detail/sexually-transmitted-infections-(stis)